CLINICAL TRIAL: NCT05012930
Title: Effects of Complementary Feeding on Infant Growth and Gut Health
Acronym: MINT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 20-2232; 1R01DK126710-01 (NIH)
Record Dates: First submitted 2021-08-12; First posted 2021-08-19 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Gut Microbiome; Linear Growth

STUDY DESIGN:
Intervention Model Description: 6 months intervention from ~5-12 months with follow-up assessments at 18 and 24 months.
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Study Provided Diet - Meat (Experimental): A group of complementary foods provided to participants by researchers.
  Interventions: Other: Baby Foods - Meat
- Study Provided Diet - Plant (Experimental): A group of complementary foods provided to participants by researchers.
  Interventions: Other: Baby Foods - Dairy
- Study Provided Diet - Dairy (Experimental): A group of complementary foods provided to participants by researchers.
  Interventions: Other: Baby Foods - Plant
- Traditional Diet (Placebo Comparator): No study foods provided to participants by researchers. Participants will eat a typical diet provided by caregivers.
  Interventions: Other: Foods from the home

INTERVENTIONS:
Other: Baby Foods - Meat — Commercially available baby foods
  Arms: Study Provided Diet - Meat
Other: Baby Foods - Dairy — Commercially available baby foods
  Arms: Study Provided Diet - Plant
Other: Baby Foods - Plant — Commercially available baby foods
  Arms: Study Provided Diet - Dairy
Other: Foods from the home — Caregiver will provide participant with usual foods from the home
  Arms: Traditional Diet

SUMMARY:
This study plans to learn more about how consuming different foods during the time of early complementary feeding (~5 to 12 months) affects growth and the development of bacteria living inside your baby's gut through school-age. The results from this study will potentially help to support future recommendations and dietary guidance for infant feeding practices.

The three primary aims include:

Aim 1. Identify the impact of dietary patterns with different protein-rich foods on infant growth.

Aim 2. Identify the impact of dietary patterns with different protein-rich foods on infant gut microbiota development.

Aim 3. Identify gut microbial taxa and genes that affect infant growth.

DETAILED DESCRIPTION:
Some details are intentionally left to out to preserve the scientific integrity of the study, and they will be included in the record after the study is completed.

ELIGIBILITY:
Inclusion Criteria:

* Full term;
* Generally healthy without conditions that would affect protein metabolism or growth
* No previous complementary food exposure
* Vaginal delivery
* No prior exposure of antibiotics during delivery or after birth
* Able to consume study foods
* Single birth.

Exclusion Criteria:

* Pre-term infants.
* Having conditions that would affect normal growth
* Had complementary foods prior to the start of the study
* Not willing to consume the complementary foods provided
* Antibiotics exposure during delivery or from birth to 5 months of life
* Multiple births

Ages: 4 Months to 60 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 267 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2025-08-01 (Actual); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Weight | Over 6 months
  Measured in kg
Length | Over 6 months
  Measured in cm
Body composition | Over 6 months
  Body fat mass, fat-free mass measured by stable isotopes
Gut Microbiome | Over 6 months
  Gut microbiota structure by 16S sequencing

SECONDARY OUTCOMES:
Total calories in breast milk | Over 6 months
  Measured in kcal/100 mL
Total carbohydrates in breast milk | Over 6 months
  Measured in g/100 mL
Total protein in breast milk | Over 6 months
  Measured in g/100 mL
Total fat in breast milk | Over 6 months
  Measured in g/100 mL
Serum IGF-1 (Insulin-like growth factor1/ somatomedin C) | Over 6 months
  Measured in ng/mL
Serum IGFBP-3 (Insulin-like growth factor-binding protein 3) | Over 6 months
  Measured in ng/mL
Serum c-reactive protein (CRP-hs) | Over 6 months
  Measured in mg/L
Plasma alpha 1-acid glycoprotein (AGP) | Over 6 months
  Measured in mg/L
Dietary intake | Over 6 months
  3 day dietary recall with results generated by NDSR software
Food acceptance | Over 6 months
  Coded from behavioral observations and consumption measured in g

CONTACTS AND LOCATIONS:
Locations (1):
- University of Colorado Anschutz Medical Campus, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tang M, Matz KL, Berman LM, Davis KN, Melanson EL, Frank DN, Hendricks AE, Krebs NF. Effects of Complementary Feeding With Different Protein-Rich Foods on Infant Growth and Gut Health: Study Protocol. Front Pediatr. 2022 Jan 13;9:793215. doi: 10.3389/fped.2021.793215. eCollection 2021. PMID 35096709